CLINICAL TRIAL: NCT00688194
Title: Overcoming Endocrine Resistance in Metastatic Breast Cancer: A Randomized Trial With Factorial Design Comparing Fulvestrant ± Lapatinib ± Aromatase Inhibitor in Metastatic Breast Cancer Progressing After Aromatase Inhibitor Therapy
Brief Title: Fulvestrant With or Without Lapatinib and/or Aromatase Inhibitor Therapy in Treating Postmenopausal Women With Metastatic Breast Cancer That Progressed After Previous Aromatase Inhibitor Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Mammella (GIM) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000596572; GIM-GIM8-OVER; EUDRACT-2007-006031-30; EU-20853; GSK-GIM-GIM8-OVER; ZENECA-GIM-GIM8-OVER
Record Dates: First submitted 2008-05-30; First posted 2008-06-02 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Fulvestrant; Lapatinib; Letrozole

ARMS (4):
- Arm I (Active Comparator): Patients receive fulvestrant intramuscularly (IM) on days 0, 14, and 28 of course 1 and on day 1 of all subsequent courses. Patients also receive oral placebo once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fulvestrant; Other: placebo
- Arm II (Active Comparator): Patients receive fulvestrant and placebo as in arm I. Patients also receive aromatase inhibitor (AI) therapy (e.g., exemestane, anastrozole, or letrozole) according to standard treatment regulations.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: fulvestrant; Drug: letrozole; Other: placebo
- Arm III (Active Comparator): Patients receive fulvestrant as in arm I and oral lapatinib tosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fulvestrant; Drug: lapatinib ditosylate
- Arm IV (Active Comparator): Patients receive fulvestrant as in arm I and lapatinib as in arm III. Patients also receive AI therapy according to standard treatment regulations.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: fulvestrant; Drug: lapatinib ditosylate; Drug: letrozole

INTERVENTIONS:
Drug: anastrozole — Patients receive aromatase inhibitor therapy according to standard treatment regulations.
  Arms: Arm II; Arm IV
Drug: exemestane — Patients receive aromatase inhibitor therapy according to standard treatment regulations.
  Arms: Arm II; Arm IV
Drug: fulvestrant — Given intramuscularly
Drug: lapatinib ditosylate — Given orally
  Arms: Arm III; Arm IV
Drug: letrozole — Patients receive aromatase inhibitor therapy according to standard treatment regulations.
  Arms: Arm II; Arm IV
Other: placebo — Given orally
  Arms: Arm I; Arm II

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant and exemestane, anastrozole, or letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells and by lowering the amount of estrogen the body makes. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether fulvestrant is more effective with or without lapatinib and/or aromatase inhibitor therapy in treating breast cancer.

PURPOSE: This randomized phase III trial is studying fulvestrant with or without lapatinib and/or aromatase inhibitor therapy to compare how well they work in treating postmenopausal women with metastatic breast cancer that progressed after previous aromatase inhibitor therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of postmenopausal women with progressive metastatic breast cancer treated with fulvestrant with or without lapatinib tosylate and/or aromatase inhibitor therapy.

Secondary

* To compare time to progression in these patients.
* To compare overall survival of these patients.
* To compare response rates in these patients.
* To compare clinical benefit rates in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to timing of progressive disease (during adjuvant therapy vs > 12 months after completion of adjuvant therapy vs during treatment for metastatic disease). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive fulvestrant intramuscularly (IM) on days 0, 14, and 28 of course 1 and on day 1 of all subsequent courses. Patients also receive oral placebo once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive fulvestrant and placebo as in arm I. Patients also receive aromatase inhibitor (AI) therapy (e.g., exemestane, anastrozole, or letrozole) according to standard treatment regulations.
* Arm III: Patients receive fulvestrant as in arm I and oral lapatinib tosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients receive fulvestrant as in arm I and lapatinib as in arm III. Patients also receive AI therapy according to standard treatment regulations.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Metastatic disease
* Confirmed disease progression after treatment with an aromatase inhibitor (AI) administered in the adjuvant or metastatic setting

  * Must have demonstrated a prior response to AI therapy (i.e., responded after > 2 years of treatment in the adjuvant setting OR complete or partial response or stable disease after ≥ 24 weeks of treatment in the metastatic setting) AND have subsequent disease progression after completion of AI therapy
* Meets 1 of the following criteria:

  * Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral CT scan
  * Evaluable disease, defined as bone lesions, lytic or mixed (lytic and sclerotic), evaluable by plain x-ray, CT scan, or MRI

    * Lesions identified only by radionucleotide bone scan are not allowed
* No HER2/neu-overexpressing tumor (IHC 3+ or FISH+)
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive primary or metastatic tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal, as defined by any of the following criteria:

  * At least 60 years of age
  * 45 to 59 years of age and meets ≥ 1 of the following criteria:

    * Amenorrhea for ≥ 12 months and intact uterus
    * Amenorrhea for < 12 months and follicle-stimulating hormone within the postmenopausal range (including patients with hysterectomy, prior hormone replacement therapy, or chemotherapy-induced amenorrhea)

      * Patients who received prior luteinizing hormone-releasing hormone (LHRH) analogues must not have restarted their menses after cessation of therapy
  * Over 18 years of age and bilateral oophorectomy
* WHO performance status 0-2
* Life expectancy ≥ 8 months
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* LVEF normal as measured by ECHO or MUGA
* Able to swallow and retain oral medication
* No ulcerative colitis
* No malabsorption syndrome or disease significantly affecting gastrointestinal function
* No known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to fulvestrant, aromatase inhibitors, lapatinib tosylate, or excipients
* No unresolved or unstable serious toxicity from prior therapy
* No active or uncontrolled infection
* No dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* No other malignancy within the past 5 years except for adequately treated cervical carcinoma in situ, melanoma in situ, or basal cell or squamous cell carcinoma of the skin
* No other concurrent disease or condition that would make the patient inappropriate for study participation
* No serious medical disorder that would interfere with patient safety

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior radiotherapy for the primary or metastatic tumor allowed
* More than 4 months since prior LHRH analogues
* More than 30 days (or 5 half-lives, whichever is longer) since prior investigational agents
* More than 14 days since prior and no concurrent CYP3A4 inducers*, including any of the following:

  * Rifampin, rifapentine, rifabutin, or other rifamycin class agents
  * Phenytoin, carbamazepine, or barbiturates (e.g., phenobarbital)
  * Efavirenz or nevirapine
  * Oral glucocorticoids (e.g., cortisone [> 50 mg], hydrocortisone [> 40 mg], prednisone [> 10 mg], methylprednisolone [> 8 mg], or dexamethasone [> 1.5 mg])
  * Modafinil
* More than 14 days since prior and no concurrent herbal or dietary supplements*, including any of the following:

  * St. John's wort
  * Ginkgo biloba
  * Kava
  * Grape seed
  * Valerian
  * Ginseng
  * Echinacea
  * Evening primrose oil
* More than 7 days since prior and no concurrent CYP3A4 inhibitors*, including any of the following:

  * Clarithromycin, erythromycin, or troleandomycin
  * Itraconazole, ketoconazole, fluconazole (> 150 mg daily), or voriconazole
  * Delaviridine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, or lopinavir
  * Verapamil or diltiazem
  * Nefazodone or fluvoxamine
  * Cimetidine or aprepitant
  * Grapefruit or grapefruit juice
* More than 6 months since prior and no concurrent amiodarone*
* No prior fulvestrant and/or lapatinib tosylate
* No prior resection of the stomach or small bowel
* No other concurrent anticancer therapy, including chemotherapy, immunotherapy, and biologic therapy

  * Concurrent bisphosphonates allowed
* No other concurrent investigational therapy
* No concurrent participation in another clinical trial NOTE: *For patients randomized to receive lapatinib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Time to progression
Overall survival
Response rate
Clinical benefit rate

CONTACTS AND LOCATIONS:
Overall Officials: Sabino De Placido, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University Medical School, Naples, Italy